CLINICAL TRIAL: NCT07091279
Title: Randomized Controlled Trial of Propranolol for Aggression, Self-Injury, and Severe Disruptive Behavior in Adolescents and Adults With Autism
Brief Title: Propranolol for Aggression, Self-Injury, and Severe Disruptive Behavior in Adolescents and Adults With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jeremy Veenstra-vanderweele (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); New York State Institute for Basic Research (Other Government)
Responsible Party: Sponsor-Investigator, Jeremy Veenstra-vanderweele, Principal Investigator, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NYSPI2024-50; AR230160 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP), U.S. Department of Defense (DoD))
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder; Challenging Behaviour; Aggression; Severe Disruptive Behaviour Disorders; Self-injury
Keywords: autism; autism spectrum disorder; propranolol; severe disruptive behavior; aggression; challenging behavior; self-injury; randomized clinical trial; RCT; high dose propranolol; open label
MeSH Terms: conditions — Autism Spectrum Disorder; Aggression; Self-Injurious Behavior; Autistic Disorder; Problem Behavior | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propranolol (Experimental): Propranolol, oral, starting at 30 mg/day (10 mg TID), titrated weekly based on tolerability to a maximum of 600 mg/day (200 mg TID) by Week 8. Participants will remain on their highest tolerated dose for an additional 4 weeks.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Participants will receive oral placebo tablets matched in appearance and dosing schedule to Propranolol. The dose will be titrated weekly in parallel with the experimental arm, and participants will remain on the highest tolerated dose for an additional 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol, oral, titrated in weekly increments from 10 mg TID to a maximum of 200 mg TID (total daily dose: 30 mg to 600 mg at 8 weeks), based on tolerability. Participants will continue at the highest tolerated dose for additional 4 weeks. Target doses: 10 mg, 40 mg, 80 mg, 120 mg, 160 mg, 200 mg TID.
  Arms: Propranolol
Drug: Placebo — Placebo for Propranolol
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if propranolol can help reduce challenging behaviors associated with Autism Spectrum Disorder, including aggression, self-injury, and severe disruptive behaviors. Participants will be randomly assigned to receive either propranolol or a placebo (a look-alike substance that contains no drug) daily for 12 weeks. After the 12 weeks, all participants will have the opportunity to receive propranolol for an additional 12 weeks.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of high dose propranolol in 60 male and female participants between the ages of 12 and 40 years who have a diagnosis of Autism Spectrum Disorder (ASD) and experience serious challenging behaviors. Participants must meet severity criteria, defined as a Clinical Global Impression Severity (CGI-S) score of 4 or higher and an Aberrant Behavior Checklist-2 Irritability/Agitation (ABC-I/A) score greater than 18. Participants will be randomly assigned to receive either propranolol or a placebo. Over the first 8 weeks, participants will gradually increase their study medication following a set schedule to find the highest dose they can tolerate (up to a maximum of 200 mg three times daily). This will be followed by 4 weeks at a steady dose. After completing the 12-week randomized phase, participants will be offered the option to learn their group assignment (propranolol or placebo) and continue into a 12-week open-label extension, where all participants will receive propranolol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-40 years.
* Clinical best-estimate diagnosis of autism spectrum disorder
* Occurrence of severe challenging behaviors, such as aggression, self-injury, and/or severely disruptive or destructive behavior, leading to safety concerns or serious impact of the quality of life, at least weekly over the past 2 months before screening.
* Score in the ASD range on the Autism Diagnostic Observation Schedule conducted at the time of study entry or in the past 5 years
* Clinical Global Impression Severity scale (CGI-S) score of 4 or above at Baseline
* Aberrant Behavior Checklist-2 Irritability/Agitation Subscale Score of 18 or above at Screening.
* A resting pulse of greater than 60 and a resting blood pressure of greater than 100/60.
* Participant must have a designated study partner who spends a minimum of 5 hours/week with the participant, and can, in the opinion of the investigator, provide a reliable report on the participant's behaviors, symptoms, and complete or supervise at-home safety monitoring and other assessments required during the study
* Participants of childbearing potential who are sexually active must agree to practice effective contraception from time of screening through 30 days after their last dose of study drug. Effective contraception is the use of two methods of contraception: hormonal contraceptives or intrauterine device and barrier (i.e., condoms, diaphragm, or cervical cap).
* Participant must be able to fully swallow study medication capsule.
* English must be primary language for participant. Study partner must be able to consent in English and complete study related form in English.

Exclusion Criteria:

* Those who are unable to provide informed consent and have no parent/guardian/legally authorized representative to provide informed consent for study enrollment
* Change in psychotropic medication or behavioral intervention (except when caused by vocational, habilitation, or school schedule) within two months before randomization.
* Asthma or history of any disorder involving bronchoconstriction in the past 5 years.
* Cardiovascular history in which the use of propranolol at high doses would be contraindicated, as determined by consulting cardiologist (such as AV block, sick sinus syndrome, valvular pathologies, cardiomyopathies, or vascular disease).
* Uncontrolled seizure disorder (a seizure within the past year and/or changes in seizure medication in the previous six months).
* Diabetes mellitus
* History of lactose intolerance that requires the potential participant to abstain from all dairy products or to take lactase supplements.
* Medical history of renal or hepatic impairment.
* Medical history of hypoglycemia
* Inability to provide blood testing when there is a medical indication for blood testing to allow clinical safety determination by the study safety physician
* Depressive episode currently or within the previous six months
* History of allergy or adverse reaction to propranolol or another beta-blocker
* Current use of any of the following: propafenone, quinidine, amiodarone, lidocaine, digitalis glycosides, calcium channel blockers, ACE inhibitors, clonidine, alpha blockers, reserpine, inotropic agents (epinephrine), isoproterenol and dobutamine, nonsteroidal anti-inflammatory drugs (indomethacin), antidepressants (MAO inhibitors, tricyclics), anesthetic agents (methoxyflurane, trichloroethylene), warfarin, neuroleptics (haloperidol), thyroxine, alcohol
* Any other medical disorder or medication which would contraindicate the use of propranolol.
* Is judged to be inappropriate for the study for any reason by the Investigator
* Has recently participated in another investigational medication study or device study within last 3 months
* Participant is unable to complete blood pressure or ECG safety assessments
* If female, is pregnant or breastfeeding.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of safety concerns and side effects associated with high-dose propranolol, including changes in blood pressure, pulse, and occurrence of dysrhythmias. | From baseline through end of treatment phase at 12 weeks
  Any participant reported side effects or adverse events will be monitored through weekly medical monitoring visits with the study safety physician. Participants will complete blinded home monitoring of blood pressure and pulse on the first three days each dosing week (baseline through end of treatment phase at 12 weeks), and pre- and post-intervention Holter monitoring will be completed for dysrhythmias (at screening and week 6)

SECONDARY OUTCOMES:
Evaluate propranolol for the treatment of severe behaviors in autistic adolescents and adults | Every 2 weeks from baseline through the end of the treatment phase at 12 weeks
  Assessed using the Aberrant Behavior Checklist-Community (ABC-C) Irritability/Agitation Subscale. The ABC-C is a global behavior checklist that measures drug and other treatment effects in people with developmental disabilities. It is made up of five subscales, including Irritability, Lethargy, Inappropriate Speech, Hyperactivity, and Stereotypy based on 58 items that describe various behavioral problems.
  The Irritability/Agitation Subscale (15-item questionnaire) will serve as the primary dependent measure. Each item is rated on a 4-point Likert scale, ranging from 0 (not a problem) to 3 (severe problem). The scores will range from minimum value of 0 to maximum value of 45, with higher score indicating worse outcome. The scale will be rated every 2 weeks from baseline to end of treatment phase.

OTHER OUTCOMES:
To test whether those with a functional explanation for severe behaviors will respond to propranolol similarly to those with less evidence of functionally based behavior. | Every 4 weeks from baseline through the end of the treatment phase at 12 weeks
  We hypothesize that participants who demonstrate greater environmentally mediated function(s) on the Questions about Behavior Function scale (QABF) scale will benefit less from propranolol. The QABF is an indirect assessment of behavioral function for individuals with developmental disabilities. It contains 25 items. The QABF yields five behavioral function categories: Access to Attention, Escape from Demands, Physical, Access to Tangible, and Nonsocial. Each question is scored with frequency descriptors of Never=0, Rarely=1, Some=2, and Often=3. Subscale scores can range from minimum value of 0 to maximum value of 15, with higher scores indicating a stronger influence of that specific behavioral function in maintaining the challenging behavior. The QABF will be administered every 4 weeks to examine whether challenging behavior serves a specific function and if so, examine whether propranolol potentially changes the function or the strength of those functions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Veenstra-VanderWeele, MD, Principal Investigator — New York State Psychiatric Institute; Eric London, MD, Principal Investigator — New York State Institute for Basic Research (IBR)
Locations (2):
- United States (2):
  - New York State Institute for Basic Research (IBR), Staten Island, New York
  - Center for Autism and the Developing Brain, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be submitted to the NIMH Data Archive (NDA). NDA is a computer system run by the National Institute of Mental Health (NIMH) that allows researchers to collect and share information with each other. During and after the study, the researchers will send health and behavioral information about the subject, in some cases, the subject's genetic information, to NDA. However, before they send it to NDA, names, addresses, phone numbers, and other identifiable information will be removed, and replaced that information with a code number called a Global Unique Identifier (GUID). Other researchers nationwide can then file an application with the National Institutes of Health to obtain access to this study data for research purposes.
Supporting Information: CSR
Access Criteria: Only approved researchers with NDA access will be able to use the data